CLINICAL TRIAL: NCT03784885
Title: A Phase 2, Double-blind, Randomized Controlled Study to Evaluate Immunogenicity and Safety of Intranasal Trivalent Influenza Virus Vaccine in Healthy Adult V Olunteers
Brief Title: A Phase 2, Double-blind Study to Evaluate Intranasal Trivalent Influenza Virus Vaccine in Healthy Adult
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1066021486
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Influenza Infection
Keywords: adjuvant; vaccine; mucosa; IgA; Escherichia coli Enterotoxin
MeSH Terms: interventions — heat-labile enterotoxin, E coli

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 μg of AD07010 (Experimental): All subjects in this group received 2 doses of 22.2 μg HA antigens from inactivated trivalent influenza vaccine in 30 μg of AD07010
  Interventions: Biological: AD07010; Biological: Inactivated trivalent influenza vaccine
- 45 μg of AD07010 (Experimental): All subjects in this group received 2 doses of 22.2 μg HA antigens from inactivated trivalent influenza vaccine in 45 μg of AD07010
  Interventions: Biological: AD07010; Biological: Inactivated trivalent influenza vaccine
- AD07010 (Active Comparator): All subjects in this group received 2 doses of 22.2 μg HA antigens from inactivated trivalent influenza vaccine
  Interventions: Biological: Inactivated trivalent influenza vaccine

INTERVENTIONS:
Biological: AD07010 — A protein based adjuvant
  Other Names: LTh(αK); Escherichia coli heat-labile enterotoxin
  Arms: 30 μg of AD07010; 45 μg of AD07010
Biological: Inactivated trivalent influenza vaccine — Inactivated trivalent seasonal influenza vaccine

SUMMARY:
The objectives of this phase 2 study are to evaluate immunogenicity, safety and tolerability of AD07030, a trivalent influenza virus antigens vaccine, given intranasally in 2 doses in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a Phase 2 prospective, randomized controlled, double-blind, multi-center study to evaluate the immunogenicity, safety and tolerability of AD07030, a trivalent influenza virus antigens vaccine, given intranasally in healthy adult volunteers.

About 358 healthy subjects, meeting all the eligibility criteria will be enrolled into the study and randomized into 3 study groups (in 2:2:1 ratio) to receive either the study vaccine at one of the dose levels of adjuvant AD07010 (30μg or 45μg LTh(αK)) in combination with hemagglutinin (HA) antigens or to receive control vaccine consisting of HA antigens alone. The 3 study groups are as follows:

* Group 1: 22.5μg HA with 30μg AD07010
* Group 2: 22.5μg HA with 45μg AD07010
* Group 3: 22.5μg HA alone Each subject will receive intranasal administration of 2 doses of IP (study or control vaccine) at same dosages, given 7 days apart on study Day 1 and Day 8. Solicited local and general AEs will be recorded after each vaccination in the subject's diary card for up to 7 days (the vaccine administration day and 6 days following it). Subjects will be followed up for monitoring of safety and immunogenicity for 180 days. AE and SAE and concomitant medication/vaccination will be collected throughout the study. There will be total of 6 study visits and a telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects aged between 20-70 (included) years.
* Should be physically and mentally healthy and free of significant medical condition as determined by Medical history, Physical examination and Clinical judgment of the Investigator.
* Negative urine β-human chorionic gonadotropin in women of childbearing potential (WOCBP; defined as women ≤ 50 years old of age or history of amenorrhea for ≤12 months) prior to administration of first dose of Investigational Product.
* WOCBP and male subjects having female partners, who are WOCBP, should be protected by effective contraceptive method (e.g. oral contraceptive and condom, intra- uterine device and condom, diaphragm with spermicide and condom) throughout the study period.
* Willing and able to give written informed consent prior to Screening and comply with study procedure.

Exclusion Criteria:

* Received vaccination against influenza within 6 months prior to Screening.
* Received any vaccination (other than influenza) within 28 days prior to Screening.
* Has previously experienced anaphylaxis or a life-threatening reaction; or has history of allergy or hypersensitivity to egg proteins, chicken proteins, any of the components of Investigational Product, or other vaccine containing same substances.
* History of influenza infection (confirmed either clinically, serologically or microbiologically) within the 6 months prior to administration of first dose of Investigational Product.
* Had active allergic rhinitis within 28 days prior to administration of first dose of Investigational Product.
* Has documented history of diarrhea within 28 days prior to administration of first dose of Investigational Product.
* Have used or been administered any intranasal medication or nasal topical treatment within 7 days prior to Screening.
* Acute respiratory illness within 7 days prior to administration of first dose of Investigational Product.
* Had administration of systemic antibiotics or antivirals within 7 days prior to Screening (excluding topical/external use of antibiotics).
* Acute sinusitis or chronic sinusitis accompanying acute symptoms within 3 days prior to administration of first dose of Investigational Product.
* With acute disease (defined as fever with body temperature >38.0°C), within 3 days prior to administration of first dose of Investigational Product.
* Having any serious chronic illness, including but not limited to, cardiovascular, pulmonary, hepatic, metabolic, renal or any auto-immune disorders, at a stage that could interfere with trial conduct or completion.
* Any confirmed or suspected immunosuppressive or immune-deficient condition, based on medical history and physical examination.
* Documented history of Bell's palsy or neurological disorder.
* Receive aspirin (Salicylate) anytime in the study from screening (Visit 1)
* A positive test for HIV antibody
* Receipt of any immunoglobulins and/or blood products within 3 months of study Screening.
* Pregnant or breast-feeding women
* Require extended long-term use of steroids including parenteral steroids or high dose inhaled steroids or have used within 28 days prior to Screening
* Participated in any other clinical investigation or use of any investigational therapy other than AD07030, within 4 weeks (28 days) or 5 half-lives, whichever is longer, before Screening.
* Unable to communicate reliably with the Investigator or unlikely to cooperate with the requirements of the study procedures or schedule, or other cases judged by the Investigator to be ineligible for participation in the study.
* Other cases judged by the Investigator to be ineligible for participation in the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-07 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer changes on Day 29 | 29 days
  Change from pre- to post-vaccination serum Geometric mean titers (GMT) of hemagglutinin inhibition (HI) antibody at Day 29(±2)

SECONDARY OUTCOMES:
Immunogenicity (HI titers) | 29, 90 and 180 days
  Derived variables: in terms of HI titers for: Seroconversion Rate (SCR), Seroconversion Factor (SCF), and Seroprotection Rate (SPR)
Immunogenicity (IgA titers) | 29, 90 and 180 days
  Change from pre- to post-vaccination GMT of mucosal anti-HA IgA antibody
Immunogenicity (anti-LTh(αK) antibodies) | 29, 90 and 180 days
  Change from pre- to post-vaccination GMT of anti- LTh(αK) antibodies
Viral neutralization | 29, 90 and 180 days
  Change from pre- to post-vaccination GMT of virus neutralization titer

CONTACTS AND LOCATIONS:
Locations (1):
- Advagene Biopharma, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pan SC, Hsu WT, Lee WS, Wang NC, Chen TJ, Liu MC, Pai HC, Hsu YS, Chang M, Hsieh SM. A double-blind, randomized controlled trial to evaluate the safety and immunogenicity of an intranasally administered trivalent inactivated influenza vaccine with the adjuvant LTh(alphaK): A phase II study. Vaccine. 2020 Jan 29;38(5):1048-1056. doi: 10.1016/j.vaccine.2019.11.047. Epub 2019 Dec 4. PMID 31812463